CLINICAL TRIAL: NCT00425490
Title: Phase III Study on the Effect of Sitagliptin on Maximal Beta Cell Stimulation
Brief Title: Effect of Januvia on Beta Cell Function in Patients With Diabetes Mellitus
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sheba Medical Center (Other Government)
Responsible Party: Ohad Cohen, Sheba medical center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SHEBA-06-4373-OC-CTIL
Record Dates: First submitted 2007-01-22; First posted 2007-01-23 (Estimated); Last update posted 2009-09-23 (Estimated); Status verified 2009-09

CONDITIONS: Diabetes Mellitus Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Sitagliptin Phosphate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: sitagliptin

SUMMARY:
The study is designed to investigate the effect of 18 weeks treatment with Sitagliptin 100 mg/day on the insulin secretion capacity of beta cells.

Patients who meet the study enrollment criteria will undergo 2 experiments (see description below); a graded hyperglycemic technique and a meal test, prior to randomization and after a 12-wk double-blind study period. The treatment effect will shed light on the magnitude of the beta cell capacity to increase its mass and function.

DETAILED DESCRIPTION:
Study design and duration: This will be an Israeli three center study. Study drug: Sitagliptin 100 mg. The study will be a double blind, randomized two arms parallel group study. The duration of the study will be up to 18 weeks (with 8 visits) for each patient. This will include: a screening period of up to 4 weeks (Visit 1 to visit 2), a 2 week single blind, placebo run-in period (visit 2 to visit 4), and a 12 week placebo controlled, double blind treatment period (visit 4 to visit 8).

Patients with T2DM who have not been treated with an AHA, or who are on AHA monotherapy or low dose oral combination therapy (low dose defined as ≤50% of the maximum labeled dose of each agent), may participate if they meet all enrollment criteria. Patients eligible to be randomized will have a HbA1c ³6.5% and £10% .

Patients who meet the study enrollment criteria will undergo 2 experiments (see description below); a graded hyperglycemic technique and a meal test, prior to randomization (Visit 3 and 4). These experiments will be will be completed after a 12-hour overnight fast. The 2 experiments will be repeated at the conclusion of the 12-wk double-blind study period (Visits 7 and 8).

Efficacy measurements: (1) Glycemic control : FPG, HbA1c, β-cell Function Parameters(Φs, Φd, Φb, Φ, Φob, T), Insulin Secretion Rate (determined from C-peptide deconvolution), 1st and 2nd phase insulin secretion, Insulin response after arginine injection, Insulin sensitivity index, glucose, insulin, C-peptide total and incremental area under the curve.

ELIGIBILITY:
Inclusion criteria:

* Patient has T2DM diagnosed within the past 5 years
* Patient is >18 and <65 years of age
* Patient is not pregnant, breast feeding and unlikely to conceive
* Patient understands the study procedures, and agrees to participate in the study by giving written informed consent
* Patient meets one of the following criteria:

  1. Patient is currently not on an AHA and has a Visit 1 HbA1c ≥6.5% and ≤10%. OR
  2. Patient is currently on AHA monotherapy or low dose (i.e. ≤50% maximum labeled dose of each agent) oral combination therapy and has a Screening/Visit 1 HbA1c ≥6.5% and ≤9.5%.
* At visit 2, patient has a HbA1c of ≥6.5% and ≤10%

Exclusion Criteria:

* Patient has type 1 diabetes mellitus
* Patient required insulin therapy within 12 weeks of Visit 1. Note: patients who received a brief period of insulin treatment (e.g., several days during a hospitalization) and who are no longer requiring insulin treatment may participate
* Patient is currently or within 12 weeks of Visit 1 taking a TZD agent as monotherapy or in combination
* Patient is currently or within 12 weeks of Visit 1 taking Byetta.
* Patient is on corticosteroids
* Patient has a history of malignancy ≤5 years prior to signing informed consent, or >5 years without documentation of remission/cure Exception: Adequately treated basal cell or squamous cell skin cancer or in situ cervical cancer. Melanoma, leukemia, lymphoma and myeloproliferative disorders of any duration are excluded -Patient is on chemotherapy
* Patient received another investigational drug in the last 12 weeks.
* Patients with concomitant liver disease and or AST > 3 fold upper limit of normal
* Patients with kidney disease or CR>1.4 mg/dl
* Patients with anemia ( Hb <11 gr in male 10 gr in female)
* Patient with active vascular disease (coronary, peripheral or cerebrovascular)
* Patient has poorly controlled hypertension defined as systolic blood pressure >160 mm Hg or diastolic >95 mm Hg
* Proliferative retinopathy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2007-01; Primary Completion 2009-07 (Actual); Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
FPG,
HbA1c,
β-cell Function Parameters(Φs, Φd, Φb, Φ, Φob, T), Insulin Secretion Rate (determined from C-peptide deconvolution), 1st and 2nd phase insulin secretion, Insulin response after arginine injection, Insulin sensitivity index, glucose, insulin,
C-peptide total and incremental area under the curve.

CONTACTS AND LOCATIONS:
Overall Officials: Ohad Cohen, MD, Principal Investigator — Sheba Medical Center
Locations (1):
- Sheba_Medical_Center, Tel Litwinsky, Israel